CLINICAL TRIAL: NCT03612284
Title: Scleral Contact Lens Insertion Solution Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Fogt (Other)
Collaborators: Contamac Ltd (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Fogt, Associate Professor, Practice, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2017H0141
Record Dates: First submitted 2018-06-04; First posted 2018-08-02 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Irregular; Contour of Cornea
Keywords: Contact lens solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device Feasibility (Experimental): Scleral lens insertion solution study. This is not an interventional study, but a study to test a new contact lens solution. Primary FDA Classification: 21 CFR 886.5928 Soft (Hydrophilic) Contact Lens Care Products Product Code: LPN
  Secondary FDA Classification: 21 CFR 886.5918 - Rigid gas permeable contact lens care products Product Code: MRC
  The FDA has previously made risk determinations (class II, non-significant risk) for devices classified under 21 CFR 886.5928 and 21 CFR 886.5918. As a non-significant risk device, the GatorFil Contact Lens Saline Solution is exempt from the IDE regulation (21 CFR 812).
  Interventions: Device: contact lens insertion solution

INTERVENTIONS:
Device: contact lens insertion solution — This contact lens solution is being tested for safety and comfort and is not an "intervention." Subjects will have their scleral contact lenses filled with the test saline in the examination room and applied to their eyes. They will be monitored for symptoms and will be examined. Six to 8 hours later or whenever their lens clouding typically occurs they will return for further assessment and dispensing of solution if acceptable. subjects will use the solution for 5-9 days and return for a follow-up appointment. At each visit, subjects will complete an OSDI questionnaire and a Current Symptoms questionnaire.

SUMMARY:
The purpose of this study is to determine the clinical ocular compatibility (feasibility of safety and efficacy) of a patented solution (US Patent 2,259,437, Stone) which contains multiple essential ions and has a pH and tonicity which more closely mimics human tears as compared to the subjects' current habitual scleral lens insertion solution.

DETAILED DESCRIPTION:
The sterile solution is provided by prescription for each patient by a local compounding pharmacy in unit dose containers. The initial exposure - filling the posterior bowl of the scleral contact lens by the Investigator and applying the lens to the eye - will be monitored in the office for one hour, prior to any dispensing of the solution to the patient for their use at home or work.

This is a one week, unmasked comparison of the new solution to the subject's habitual solution used for scleral lens insertion. The (historical) control is the saline habitually used by the subjects.

The sample size is determined to be manageable to insure close supervision of the subjects in these initial trials and to inform us for future safety and efficacy trials.

The primary safety outcome measure will be slit lamp examination of the ocular anterior segment and the secondary outcome measure will be photo-documentation by ocular coherence tomography of the clouding of the tears between the cornea and scleral contact lens. The primary efficacy outcome will be ocular comfort as assessed by questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older.
* Wear a scleral contact lens habitually 6 or more hours a day.
* Needs to remove scleral lens due to fogging and refill or definitely reports fogging.
* Must have worn habitual scleral lens for at least 3 months
* Willing and able to attend study visits.

Exclusion Criteria:

* Currently under treatment for an eye infection or inflammation such as adapted keratoconus or healed post penetrating keratoplasty. Stable keratoconus is acceptable.
* Currently taking topical ophthalmic prescription medications.
* Current medical eye complications such as glaucoma or uveitis.
* Recent corneal surgery
* Sjogrens or other clinically significant active ocular surface disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Change in corneal staining or corneal disruption as assessed with clinical biomicroscope | immediately after first use of solution and again in 5 to 9 days
  ocular safety examination
Comfort and vision quality as assessed by Ocular Surface Disease Index (OSDI) questionnaire | 5 to 9 days
  Subjects will answer the OSDI questionnairre (score of 0-48) used to assess symptoms related to comfort and vision. The survey will be done with the subjects regular solution and repeated after using the test solution
Comfort as assessed by Current Symptoms Survey (CSS) | 5 to 9 days
  Subjects will respond to the CSS survey (scores of 0-100 for various symptoms) - used to assess symptoms related to comfort and vision. The survey will be done with the subjects regular solution and repeated after using the test solution

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Fogt, OD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No